CLINICAL TRIAL: NCT00063362
Title: Combination Therapy in Bipolar Rapid Cycling
Brief Title: Combination Therapy for the Treatment of Bipolar Disorders
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding Expiration
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Keming Gao, Director, Mood and Anxiety Clinic, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21MH062650 (NIH); R21MH062650 (NIH); DSIR AT-SO
Record Dates: First submitted 2003-06-25; First posted 2003-06-27 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-10

CONDITIONS: Bipolar Disorder
Keywords: Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lithium; Lithium Carbonate; Lamotrigine; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium + divalproex + lamotrigine (Experimental)
  Interventions: Drug: Lithium; Drug: Lamotrigine; Drug: Divalproex
- Lithium + divalproex + placebo (Placebo Comparator)
  Interventions: Drug: Lithium; Drug: Divalproex; Drug: Placebo

INTERVENTIONS:
Drug: Lithium — Lithium monotherapy was initiated at 450 mg once daily and titrated slowly over three weeks to a minimum blood level of 0.5 milliequivalent /L (mEq/L).
  Other Names: Lithium Carbonate
Drug: Lamotrigine — Patients were assigned in a one to one ratio to adjunctive lamotrigine versus placebo after stratification for illness type (bipolar I versus bipolar II), historical response to lithium (response versus non-response), and length of current exposure to combination treatment with lithium and divalproex (< 2 months versus ≥ 2 months). During Phase 2, patients were continued on the same doses of lithium and divalproex as during the open-label treatment phase and equal capsules of double-blind lamotrigine or matching placebo were gradually added per a structured dosing schedule up to a minimum dose of 150 mg and a maximum dose of 200 mg per day.
  Other Names: Lamictal
  Arms: Lithium + divalproex + lamotrigine
Drug: Divalproex — Divalproex was then initiated at 250 mg twice daily and increased slowly over five weeks to a minimum blood level of 50 μg/mL.
  Other Names: Depakote; Valproic Acid
Drug: Placebo — Patients were assigned in a one to one ratio to adjunctive lamotrigine versus placebo after stratification for illness type (bipolar I versus bipolar II), historical response to lithium (response versus non-response), and length of current exposure to combination treatment with lithium and divalproex (< 2 months versus ≥ 2 months). During Phase 2, patients were continued on the same doses of lithium and divalproex as during the open-label treatment phase and equal capsules of double-blind lamotrigine or matching placebo were gradually added per a structured dosing schedule up to a minimum dose of 150 mg and a maximum dose of 200 mg per day.
  Arms: Lithium + divalproex + placebo

SUMMARY:
This study will compare triple and double drug regimens in the treatment of patients with depression, hypomania, or mania.

DETAILED DESCRIPTION:
Early studies have shown lithium to produce a high percentage of satisfactory clinical response in patients with bipolar disorders. These studies, however, do not include lithium-refractory subgroups, such as bipolar II disorder patients. When the wide spectrum of bipolar disorders is considered, the lithium response rate decreases significantly. More broadly effective regimens are needed.

Participants in this study will be randomly assigned to receive either lithium plus divalproex or lithium, divalproex, and lamotrigine for 7 months. Symptoms of depression and mania will be assessed with scales and patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I or II Disorder
* Meet criteria for rapid cycling, defined as four or more episodes over the past 12 months
* Meet criteria for a major depressive episode

Exclusion Criteria:

* History of intolerability of lithium, divalproex, or lamotrigine

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2002-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, MD, PhD, Principal Investigator — Case Western Reserve University / University Hospitals of Cleveland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted by the Mood Disorders Program at Case Western Reserve University/University Hospitals Case Medical Center (Cleveland, OH, USA) from August 2002 to June 2007.
Groups:
- Lithium + Divalproex + Lamotrigine: Divalproex : Divalproex was then initiated at 250 mg twice daily and increased slowly over five weeks to a minimum blood level of 50 μg/mL.
  Lamotrigine : Patients were assigned in a one to one ratio to adjunctive lamotrigine versus placebo after stratification for illness type (bipolar I versus bipolar II), historical response to lithium (response versus non-response), and length of current exposure to combination treatment with lithium and divalproex (< 2 months versus ≥ 2 months). During Phase 2, patients were continued on the same doses of lithium and divalproex as during the open-label treatment phase and equal capsules of double-blind lamotrigine or matching placebo were gradually added per a structured dosing schedule up to a minimum dose of 150 mg and a maximum.
  dose of 200 mg per day.
  Lithium : Lithium monotherapy was initiated at 450 mg once daily and titrated slowly over three weeks to a minimum blood level of 0.5 milliequivalent/L (mEq/L).
- Lithium + Divalproex + Placebo: Divalproex : Divalproex was then initiated at 250 mg twice daily and increased slowly over five weeks to a minimum blood level of 50 μg/mL.
  Lithium : Lithium monotherapy was initiated at 450 mg once daily and titrated slowly over three weeks to a minimum blood level of 0.5 mEq/L.
Period: Overall Study
Arm/Group | Lithium + Divalproex + Lamotrigine | Lithium + Divalproex + Placebo
Started | 23 | 26
Completed | 19 | 22
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Lithium + Divalproex + Lamotrigine: Divalproex : Divalproex was then initiated at 250 mg twice daily and increased slowly over five weeks to a minimum blood level of 50 μg/mL.
  Lamotrigine : Patients were assigned in a one to one ratio to adjunctive lamotrigine versus placebo after stratification for illness type (bipolar I versus bipolar II), historical response to lithium (response versus non-response), and length of current exposure to combination treatment with lithium and divalproex (< 2 months versus ≥ 2 months). During Phase 2, patients were continued on the same doses of lithium and divalproex as during the open-label treatment phase and equal capsules of double-blind lamotrigine or matching placebo were gradually added per a structured dosing schedule up to a minimum dose of 150 mg and a maximum.
  dose of 200 mg per day.
  Lithium : Lithium monotherapy was initiated at 450 mg once daily and titrated slowly over three weeks to a minimum blood level of 0.5 mEq/L.
- Total: Total of all reporting groups
Arm/Group | Lithium + Divalproex + Lamotrigine | Lithium + Divalproex + Placebo | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (11.0) | 43.0 (9.6) | 37.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 21 | 24 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Bipolar Subtype [Number; unit: participants] — Bipolar I Disorder is mainly defined by manic or mixed episodes that last at least seven days, or by manic symptoms that are so severe that the person needs immediate hospital care.
  Bipolar II Disorder is defined by a pattern of depressive episodes shifting back and forth with hypomanic episodes, but no full manic or mixed episodes
  participants
    Bipolar I disorder | 11 | 16 | 27
    Bipolar II disorder | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Experience a Marked and Persistent Bimodal Response
Description: A marked bimodal response is defined by the following three conditions over four consecutive weeks while on triple therapy and after three weeks of ltg:
  1. Montgomery Asberg Depression Rating Scale (MADRS) total score of <= 19
  2. Young Mania Rating Scale (YMRS) total score of <= 12.5
  3. Global Assessment Scale (GAS) score >= 51
  The MADRS measures the severity of a subject's depression symptoms with a possible total score ranging from 0 - 60, with higher scores indicating more severe depression.
  The YMRS measures the severity of a subject's manic symptoms with a possible total score ranging from 0 - 60, with higher scores indicating more severe mania.
  The GAS measures a used to rate subjectively the social, occupational, and psychological functioning of a subject and ranges in score from 0-100, with a higher score indicating better social, occupational, and psychological functioning.
Time Frame: Baseline and Week 28
Measure: Number; unit: participants
Arm/Group | Lithium + Divalproex + Lamotrigine | Lithium + Divalproex + Placebo
Number analyzed (Participants) | 23 | 26
participants | 7 | 8

ADVERSE EVENTS:
Arm/Group | Lithium + Divalproex + Lamotrigine | Lithium + Divalproex + Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 2/23 | 1/26
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium + Divalproex + Lamotrigine (N=23) | Lithium + Divalproex + Placebo (N=26)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes